CLINICAL TRIAL: NCT01754337
Title: An Open-label, Randomized, Three-way, Cross-over Study to Assess the Efficacy of Single-hormone Closed-loop Strategy, Dual-hormone Closed-loop Strategy and Conventional Pump Therapy in Regulating Glucose Levels During 24 Hours in Adults and Adolescents With Type 1 Diabetes
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) for 24 Hours in Adults and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: McGill University (Other); Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-03
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia; Insulin; Glucagon; Closed-loop system; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single-hormone closed-loop system (Active Comparator): In single-hormone closed-loop system, variable subcutaneous insulin infusion rate will be used to regulate glucose levels.
  Interventions: Other: Closed-loop system
- Dual-hormone closed-loop system (Active Comparator): In dual-hormone closed-loop system, variable subcutaneous insulin and glucagon infusion rates will be used to regulate glucose levels.
  Interventions: Other: Closed-loop system
- Insulin pump therapy (Active Comparator): Patient's conventional treatment will be implemented.
  Interventions: Other: Closed-loop system

INTERVENTIONS:
Other: Closed-loop system — Patients will be admitted at the research clinical facility at 7:00. At 8:00, a mixed meal will be served. At 9:00, patients will be asked to perform two 30-min standardized activities. At 12:00, a mixed meal will be served. At 13:00, patients will be asked to perform two 30-min activities. At 17:00, a mixed meal will be served. At 19:30, patients will perform 60 minutes of aerobic treadmill exercise at an intensity of 60% VO2max. A bedtime snack of 20g carbohydrate will be given at 21:00. Patients will be discharged at 8:00 the next morning

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormone: insulin and glucagon.

The main objective of this project is to compare the efficacy of single-hormone closed-loop strategy, dual-hormone closed-loop strategy and pump therapy to regulate glucose levels in a 24-hours in-patient study with standardized conditions in adults and adolescents with type 1 diabetes.

The investigators hypothesized that dual-hormone closed-loop strategy is more effective in regulating glucose levels in adults and adolescents with type 1 diabetes compared to single-hormone closed-loop strategy, which in turn is more effective than the conventional pump therapy.

DETAILED DESCRIPTION:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosages based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormone: insulin and glucagon.

We aim to conduct the 1st randomized three-way cross-over trial comparing single hormone closed-loop strategy, dual-hormone closed-loop strategy and the conventional pump therapy. We aim to compare the three interventions for 24 hours in adults and adolescents with type 1 diabetes. Each 24 hours will include a 60-min exercise session, three meals characterizing a full day, activities that mimick real-life conditions and an overnight stay. This study will also allow for multiple comparisons and evaluating the benefits of each component separately (i.e. the benefits of merely closing the loop with insulin alone vs. adding glucagon to the closed-loop strategy).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 12 years of old.
2. Clinical diagnosis of type 1 diabetes for at least one year. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. HbA1c ≤ 12%.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. A recent injury to body or limb, muscular disorder, use of any medication or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol.
4. Pregnancy.
5. Severe hypoglycemic episode within two weeks of screening.
6. Current use of glucocorticoid medication (except low stable dose).
7. Known or suspected allergy to the trial products or meal contents.
8. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
9. Anticipating a significant change in exercise regimen between admissions (i.e. starting or stopping an organized sport).
10. Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percentage of time of plasma glucose levels spent in target range. | 24 hours
  Two-hour postprandial target range is between 4.0 and 10.0 mmol/l. Otherwise, target range is defined to be between 4.0 and 8.0 mmol/l.

SECONDARY OUTCOMES:
Percentage of time of plasma glucose levels spent in the low range | 24 hours
  Low range is defined to be a. below 4 mmol/L; b. below 3.5 mmol/L; c. below 3.3 mmol/L.
Percentage of overnight time of plasma glucose levels spent in the low range | 9 hours
  Low range is defined to be a. < 4 mmol/L; b. < 3.5 mmol/L; c. < 3.3 mmol/L.
Standard deviation of glucose levels | 24 hours
  Measure of glucose variability
Total insulin delivery | 24 hours
Mean plasma glucose level | 24 hours
Mean plasma glucose level | 9 hours
Mean plasma insulin concentration | 24 hours
Mean plasma glucagon concentration | 24 hours
Number of subjects experiencing hypoglycemia requiring oral treatment | 24 hours
  Number of subjects experiencing hypoglycemia requiring oral treatment during a. the overall study period; b. the exercise; c. the night.
Percentage of time of plasma glucose levels spent between 4.0 and 10.0 mmol/L | 24 hours
Percentage of overnight time of plasma glucose levels spent between 4.0 and 8.0 mmol/L | 9 hours
Percentage of overnight time of plasma glucose levels spent between 4.0 and 10.0 mmol/L | 9 hours
Percentage of time of plasma glucose levels spent in the high range | 24 hours
  High range is defined to be above a. 8.0 mmol/L; b. 10.0 mmol/L
Percentage of overnight time of plasma glucose levels spent in the high range | 9 hours
  High range is defined to be above a. 8.0 mmol/L; b. 10.0 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Haidar A, Legault L, Messier V, Mitre TM, Leroux C, Rabasa-Lhoret R. Comparison of dual-hormone artificial pancreas, single-hormone artificial pancreas, and conventional insulin pump therapy for glycaemic control in patients with type 1 diabetes: an open-label randomised controlled crossover trial. Lancet Diabetes Endocrinol. 2015 Jan;3(1):17-26. doi: 10.1016/S2213-8587(14)70226-8. Epub 2014 Nov 27. PMID 25434967